CLINICAL TRIAL: NCT01103414
Title: Phase 2B, Randomized, Double-Blind, Comparator- & Placebo-Controlled, Dose Ranging Study to Evaluate Safety, Tolerability & Efficacy of 3 Dose Levels of Mitoglitazone in Type 2 Diabetic Patients
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of Three Dose Levels of Mitoglitazone in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metabolic Solutions Development Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSDC-C004
Record Dates: First submitted 2010-04-07; First posted 2010-04-14 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — MSDC-0160; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Mitoglitazone 50 mg capsules (Experimental): Mitoglitazone 50 mg capsules self administered once-daily each morning after an overnight fast and 30 minutes before the morning meal for 84 days.
  Interventions: Drug: Mitoglitazone
- Mitoglitazone 100 mg capsules (Experimental): Mitoglitazone 100 mg capsules self administered once-daily each morning after an overnight fast and 30 minutes before the morning meal for 84 days.
  Interventions: Drug: Mitoglitazone
- Mitoglitazone 150 mg capsules (Experimental): Mitoglitazone 150 mg capsules self administered once-daily each morning after an overnight fast and 30 minutes before the morning meal for 84 days.
  Interventions: Drug: Mitoglitazone
- Pioglitazone 45 mg capsules (Active Comparator): Pioglitazone 45 mg capsules self administered once-daily each morning after an overnight fast and 30 minutes before the morning meal for 84 days.
  Interventions: Drug: Pioglitazone
- Matching placebo (Placebo Comparator): Placebo capsules self administered once-daily each morning after an overnight fast and 30 minutes before the morning meal for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mitoglitazone — 50 mg capsules, once daily for 84 days
  Other Names: MSDC-0160
  Arms: Mitoglitazone 50 mg capsules
Drug: Mitoglitazone — Mitoglitazone 100 mg capsules, once daily for 84 days
  Other Names: MSDC-0160
  Arms: Mitoglitazone 100 mg capsules
Drug: Mitoglitazone — Mitoglitazone 150 mg capsules, once daily for 84 days
  Other Names: MSDC-0160
  Arms: Mitoglitazone 150 mg capsules
Drug: Pioglitazone — Pioglitazone 45 mg, once daily for 84 days
  Other Names: ACTOS
  Arms: Pioglitazone 45 mg capsules
Drug: Placebo — Placebo, once daily for 84 days
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of three dose levels of Mitoglitazone™ (MSDC-0160) in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The primary study objectives are to characterize the reduction in fasting plasma glucose in response to three different doses of Mitoglitazone as compared to placebo following once-daily dosing for 84 consecutive days (12 weeks) in patients with Type 2 diabetes and to investigate the safety and tolerability of three different doses of Mitoglitazone following once-daily dosing for 84 consecutive days (12 weeks) in patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria

1. Males and females with Type 2 diabetes (fasting plasma glucose ≥126 mg/dL at screening, glycosylated hemoglobin [HbA1c] >7 and ≤10%, and Insulin C-peptide >1 ng/mL). Patients can be naïve to diabetes therapy or if taking metformin should be on a stable dose level for a period of at least 3 months prior to screening visit (no dose limit).
2. Between the ages of 18-75 years, inclusive.
3. Females should be either postmenopausal (at least 12 months since last menses) or surgically sterilized (bilateral tubal ligation or hysterectomy). Menopausal status will be verified by a follicle-stimulating hormone (FSH) test. If FSH levels are below 40 mIL/mL, some method of birth control must be used. Those with bilateral tubal ligation must also use a barrier method of birth control. In addition, all females must have a negative pregnancy test at Screen and Day 15 regardless of childbearing potential. Males with female partners of child-bearing potential must agree to use adequate contraceptive methods (including a condom, plus one other form of contraception) if engaging in sexual intercourse.
4. Body Mass Index (BMI) = 23 kg/m2 to 45 kg/m2 (inclusive).
5. Willing and able to make a screening visit to the clinic and seven visits over a 21 week period.
6. Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.

Exclusion Criteria

1. Use of TZDs or diabetes medications other than metformin (generic or Glucophage®) 3 months prior to screening.
2. History of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
3. Fasting plasma glucose in excess of 240 mg/dl at screening
4. History of heart failure (including CHF) or previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 6 months prior to screening.
5. ALT and/or AST levels that are twice the upper limit of normal; bilirubin levels that exceed 2 mg/dL; serum creatinine >1.5 mg/dL in men or > 1.4 mg/dL in women.
6. History nephropathy, neuropathy, or retinopathy within 6 months of screening.
7. Use of glucocorticoids (oral, injectible, intraarticular, or chronic inhaled) or weight-loss drugs within 3 months of randomization.
8. Current or recurrent disease that may affect the action, absorption or disposition of the study treatment, or clinical or laboratory assessments.
9. Current or history of severe or unstable disorder (medical or psychiatric) requiring treatment that may make the patient unlikely to complete the study.
10. Febrile illness within the 5 days prior to the first dose.
11. Known history of HIV, hepatitis B, or hepatitis C.
12. Clinically significant findings on physical examination, including BP, pulse rate and 12-lead ECG.
13. Blood pressure greater than 160/100 mmHg. Patients with elevated BP (<160/100 mmHg) with or without current treatment will be allowed at the discretion of the Principal Investigator (PI) and primary care physician. Individuals with hypertension must have been stabilized to the current treatment regimen for at least 6 weeks prior to screening.
14. Change in BP or lipid-lowering medication within 6 weeks or change in dose of metformin or thyroid replacement within 3 months prior to screening.
15. Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds or any of their stated ingredients.
16. History of alcohol or drug abuse within 6 months of Screening.
17. Have participated in an investigational study or received an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
18. Blood donation of 1 pint or more within 56 days of screening.
19. Plasmapheresis or plasma donation within 30 days of screening.
20. Single 12-lead ECG demonstrating a QTc >450 msec at Screening. A single repeat ECG may be done at the investigator's discretion.
21. Any surgical or medical condition which may significantly alter the absorption of any drug substance including, but not limited to, any of the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active inflammatory bowel syndrome.
22. Evidence of clinically relevant pathology that could interfere with the study results or put the patient's safety at risk.
23. Malignancy, including leukemia and lymphoma (not including basal cell skin cancer) within the last 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Colca, PhD, Study Director — MSDC
Locations (24):
- United States (24):
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Chino, California
  - Los Angeles, California
  - Spring Valley, California
  - Walnut Creek, California
  - Miami, Florida
  - New Port Richley, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Grand Rapids, Michigan
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Tiffin, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Greer, South Carolina
  - Corpus Christi, Texas
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 investigational sites in the United States. Over the course of the study, 786 patients were screened, 356 patients were randomized, 297 patients completed the study, and 258 patients completed the study for the Modified Per Protocol Population which required compliance with taking the active medications.
Pre-assignment Details: The study consisted of a 14-day, placebo lead-in period & an 84-day double-blind treatment period. At screening, patients were required to have FPG ≥126 mg/dL, HbA1c 7-10%, and insulin C-peptide >1 ng/mL. At the end of the lead-in period, eligible patients were randomized based on a stratification criterion of current metformin use (yes, no).
Groups:
- Mitoglitazone 50 mg Capsules: Over-encapsulated Mitoglitazone 50 mg tablet
- Mitoglitazone 100 mg Capsules: Over-encapsulated Mitoglitazone 100 mg tablet
- Mitoglitazone 150 mg Capsules: Over-encapsulated Mitoglitazone 50 mg tablet and 100 mg tablet
- Pioglitazone 45 mg Capsules: Over-encapsulated ACTOS three 15 mg tablets
- Matching Placebo: Over-encapsulated placebo tablet
Period: Overall Study
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Started | 72 | 71 | 71 | 71 | 71
Completed | 59 | 62 | 56 | 64 | 56
Not Completed | 13 | 9 | 15 | 7 | 15

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least 1 dose of randomized study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo | Total
Number analyzed (Participants) | 72 | 71 | 71 | 71 | 71 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9.70) | 55.5 (10.19) | 56.0 (8.76) | 54.2 (9.90) | 53.4 (8.76) | 54.7 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 29 | 26 | 32 | 37 | 166
  Male | 30 | 42 | 45 | 39 | 34 | 190
Region of Enrollment [Number; unit: participants]
  United States | 72 | 71 | 71 | 71 | 71 | 356
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 176.1 (39.62) | 173.7 (36.73) | 170.2 (44.22) | 172.3 (33.96) | 170.2 (43.78) | 172.5 (39.70)
HbA1c [Mean (Standard Deviation); unit: percent] | 8.2 (0.862) | 8.09 (0.816) | 8.00 (0.809) | 8.08 (0.852) | 8.04 (0.845) | 8.08 (0.835)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12.
Description: Change from baseline in fasting plasma glucose in response to three different doses of Mitoglitazone as compared to pioglitazone following once-daily dosing for 84 consecutive days (12 weeks) in patients with Type 2 diabetes.
Time Frame: Baseline, Week 12
Population: The Modified Per-Protocol Population included all per-protocol patients (all ITT patients who completed the 12-week, double-blind treatment period without any major deviations from the protocol procedures) without any study medication non-compliance issues based on their pharmacokinetic data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 48 | 52 | 47 | 55 | 56
mg/dL | -5.3 (4.95) | -14.6 (4.74) | -25.1 (4.99) | -27.2 (4.61) | 3.8 (4.59)
Statistical Analysis 1: Comparison: Mitoglitazone 50 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p = 0.1819, ANCOVA; Mean Difference (Net) = -9.1, 95% CI 2-sided [-22.4 to 4.3], Standard Error of Mean 6.77
Statistical Analysis 2: Comparison: Mitoglitazone 100 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p = 0.0057, ANCOVA; Mean Difference (Net) = -18.4, 95% CI 2-sided [-31.4 to -5.4], Standard Error of Mean 6.59
Statistical Analysis 3: Comparison: Mitoglitazone 150 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -28.9, 95% CI 2-sided [-42.3 to -15.6], Standard Error of Mean 6.80
Statistical Analysis 4: Comparison: Pioglitazone 45 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -31.0, 95% CI 2-sided [-43.8 to -18.2], Standard Error of Mean 6.50

2. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from baseline in plasma glucose measured by hemoglobin A1c in response to three different doses of Mitoglitazone and pioglitazone as compared to placebo following once-daily dosing for 84 consecutive days (12 weeks) in patients with Type 2 diabetes.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 48 | 52 | 47 | 55 | 56
percentage of hemoglobin | -0.10 (0.129) | -0.49 (0.123) | -0.57 (0.130) | -0.69 (0.120) | 0.29 (0.119)
Statistical Analysis 1: Comparison: Mitoglitazone 50 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p = 0.0273, ANCOVA; Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.73 to -0.04], Standard Error of Mean 0.175
Statistical Analysis 2: Comparison: Mitoglitazone 100 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.13 to -0.45], Standard Error of Mean 0.171
Statistical Analysis 3: Comparison: Mitoglitazone 150 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.86, 95% CI 2-sided [-1.21 to -0.52], Standard Error of Mean 0.176
Statistical Analysis 4: Comparison: Pioglitazone 45 mg Capsules vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Net) = -0.98, 95% CI 2-sided [-1.32 to -0.65], Standard Error of Mean 0.169

3. Secondary Outcome: Percent Change From Baseline to Week 12 Endpoint in HMW Adiponectin
Description: Percent change from baseline to week 12 endpoint in high molecular weight adiponectin
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: percentage of baseline values
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 48 | 52 | 47 | 55 | 56
percentage of baseline values | 45.2 (18.15) | 94.4 (17.44) | 132.4 (18.34) | 287.0 (16.94) | 4.9 (16.82)

4. Secondary Outcome: Change From Baseline to Week 12 Endpoint in Hematocrit
Description: Change from baseline to week 12 endpoint in hematocrit as an indication of fluid retention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of volume
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 48 | 52 | 47 | 55 | 56
percentage of volume | 0.0 (0.34) | -0.9 (0.33) | -1.0 (0.34) | -1.7 (0.32) | 0.0 (0.32)

5. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Change from baseline at week 12 endpoint in hemoglobin concentration
Time Frame: 12 weeks
Population: All randomized patients who received at least 1 dose of randomized study medication and who had both baseline and week 12 assessments.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 61 | 62 | 59 | 64 | 56
g/dL | -0.07 (0.729) | -0.38 (0.720) | -0.33 (.676) | -0.60 (0.827) | -0.07 (0.670)

6. Secondary Outcome: Change From Baseline in RBC
Description: Change from baseline at week 12 endpoint in red blood cell concentration
Time Frame: 12 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10e-6 cells per uL
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 61 | 62 | 59 | 64 | 56
10e-6 cells per uL | -0.014 (0.2073) | -0.098 (0.2332) | -0.107 (0.2499) | -0.211 (0.2878) | 0.035 (0.2480)

7. Secondary Outcome: Change in Body Weight From Baseline to Week 12 Endpoint
Description: Effects of 3 different doses of Mitoglitazone and pioglitazone as compared to placebo on body weight following once-daily dosing for 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: kg
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 48 | 52 | 47 | 55 | 56
kg | 0.23 (0.318) | 0.56 (0.306) | 1.15 (0.323) | 1.53 (0.297) | -0.71 (0.294)

8. Secondary Outcome: Change From Baseline in Waist Circumference at Week 12 Endpoint
Description: Effects of 3 different doses of Mitoglitazone and pioglitazone as compared to placebo on waist circumference following once-daily dosing for 12 weeks
Time Frame: 12 weeks
Population: All randomized patients who received at least 1 dose of randomized study medication and had both baseline and week 12 waist circumference assessments
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 61 | 62 | 59 | 65 | 56
cm | 0.1 (3.39) | -0.2 (2.13) | -0.4 (4.02) | 0.7 (2.95) | -0.9 (3.21)

9. Secondary Outcome: Presence of Edema Post Baseline During 12 Weeks Active Treatment
Description: Effects of 3 different doses of Mitoglitazone and pioglitazone as compared to placebo on presence of edema following once-daily dosing for 12 weeks
Time Frame: 12 weeks
Population: All randomized patients who received at least 1 dose of randomized study medication and had both a baseline and post baseline edema assessment
Measure: Number; unit: participants
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 68 | 69 | 70 | 71 | 70
participants | 8 | 9 | 4 | 6 | 8

10. Secondary Outcome: Changes in HDL Particle Size Subfractions From Baseline to Week 12
Description: Effects of 3 different doses of Mitoglitazone and pioglitazone as compared to placebo on HDL particle size profile as characterized by changes in NMR analysis of subfractions following once-daily dosing for 12 weeks
Time Frame: 12 weeks
Population: The Modified Per-Protocol Population included all ITT patients who completed the 12-week, double-blind treatment period with no major deviations from protocol procedures, without any study medication non-compliance issues based on their pharmacokinetic data, and with both baseline and post-baseline NMR analysis of lipoprotein particle subfractions.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 43 | 48 | 45 | 51 | 56
nM | 0.00 (0.25) | 0.05 (0.40) | 0.10 (0.30) | 0.20 (0.50) | 0.00 (0.25)

11. Secondary Outcome: Changes in LDL Particle Size Subfractions From Baseline to Week 12
Description: Effects of 3 different doses of Mitoglitazone and pioglitazone as compared to placebo on LDL particle size profile as characterized by changes in NMR analysis of subfractions following once-daily dosing for 12 weeks
Time Frame: 12 week
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Number analyzed (Participants) | 43 | 48 | 45 | 51 | 56
nM | 0.20 (0.60) | 0.20 (0.55) | 0.30 (0.50) | 0.60 (0.70) | 0.00 (0.40)

ADVERSE EVENTS:
Description: The Safety Population includes all randomized subjects who received at least one dose of randomized study medication. Two subjects withdrew from the study during the placebo lead-in period.
Arm/Group | Mitoglitazone 50 mg Capsules | Mitoglitazone 100 mg Capsules | Mitoglitazone 150 mg Capsules | Pioglitazone 45 mg Capsules | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71 | 1/70 | 3/71 | 0/71
Other Adverse Events (participants affected / at risk) | 10/71 | 5/71 | 5/70 | 6/71 | 6/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitoglitazone 50 mg Capsules (N=71) | Mitoglitazone 100 mg Capsules (N=71) | Mitoglitazone 150 mg Capsules (N=70) | Pioglitazone 45 mg Capsules (N=71) | Matching Placebo (N=71)
skin laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
benign prostatic hyperplasia and calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitoglitazone 50 mg Capsules (N=71) | Mitoglitazone 100 mg Capsules (N=71) | Mitoglitazone 150 mg Capsules (N=70) | Pioglitazone 45 mg Capsules (N=71) | Matching Placebo (N=71)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Diarrhea & Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less